CLINICAL TRIAL: NCT00766727
Title: Clinical Evaluation of the GLYDe Dressing for Post-surgical Incision Care
Acronym: Mona Lisa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neodyne Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA001
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Results first posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Post Surgical Incisions From Abdominoplasty Procedures
Keywords: incision; abdominoplasty
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- GLYDe Dressing (Experimental): Investigational Dressing
  Interventions: Device: GLYDe Dressing
- Standard of Care (No Intervention): Standard of care comparator

INTERVENTIONS:
Device: GLYDe Dressing — Wound dressing intended to minimize scar formation
  Arms: GLYDe Dressing

SUMMARY:
This study will evaluate a new dressing to be used for post-incision care for abdominoplasty patients. The hypothesis is that this dressing will minimize scar formation.

DETAILED DESCRIPTION:
This study will evaluate a new dressing in up to 30 patients who have undergone an abdominoplasty procedure. They will wear the dressing through 8 weeks post surgery and the scar will be evaluated at 3 months post surgery.

ELIGIBILITY:
Inclusion Criteria:

* subjects who have undergone an abdominoplasty 1 week prior to study participation

Exclusion Criteria:

* subjects with a history of collagen vascular disease or scleroderma
* subjects with known adverse reactions to steri-strips, medical tapes or adhesives

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Longaker, MD, Study Director — Neodyne Biosciences, Inc.
Locations (1):
- Josh Korman, MD, Mountain View, California, United States

REFERENCES:
- [Derived] Gurtner GC, Dauskardt RH, Wong VW, Bhatt KA, Wu K, Vial IN, Padois K, Korman JM, Longaker MT. Improving cutaneous scar formation by controlling the mechanical environment: large animal and phase I studies. Ann Surg. 2011 Aug;254(2):217-25. doi: 10.1097/SLA.0b013e318220b159. PMID 21606834

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: The interventions provided consisted of a GLYDe dressing which was randomly assigned to the left or right side of the patient's abdomen. The opposite side of the intervention received the standard of care (SoC).
  For example, one patient wore a GLYDe Dressing on Left Side, and SoC Right Side while another patient wore GLYDe Dressing Right Side, and SoC Left Side.
Period: Overall Study
Arm/Group | All Participants
Started | 12
Completed | 9
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 39.5 [26 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Scar Evaluation at End of Treatment Period Comparing Treated to Standard of Care (Control)
Description: Professional photographs were taken 12 months postsurgery and evaluated by lay and professional panels. A 100 point Visual Analog Scale (VAS), ranging from a score of 0 for a better outcome to a score of 100 for worse outcome, will be used to assess both the Treated and Control scars at the same timepoint.
Time Frame: through 12 months
Population: Patient population undergoing elective plastic surgery.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GLYDe Dressing (Treated): The interventions provided consisted of a GLYDe dressing which was randomly assigned to the left or right side of the patient's abdomen. The opposite side of the intervention received the standard of care (SoC).
  For example, one patient wore a GLYDe Dressing on Left Side, and SoC Right Side while another patient wore GLYDe Dressing Right Side, and SoC Left Side.
- SoC (Control): Standard of care treatment group, used as the control. The opposite side of the intervention received the standard of care (SoC). For example, one patient wore a GLYDe Dressing on Left Side, and SoC on Right Side while another patient wore GLYDe Dressing Right Side, and SoC on Left Side.
Arm/Group | GLYDe Dressing (Treated) | SoC (Control)
Number analyzed (Participants) | 9 | 9
score on a scale | 18.64 (10.86) | 50.52 (15.17)
Statistical Analysis 1: Comparison: GLYDe Dressing (Treated) vs SoC (Control); Test type: Superiority; Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -31.88, Standard Deviation 14.25

ADVERSE EVENTS:
Time Frame: 6 months
Description: The incidence and severity of wound related adverse events and infections will be summarized and compared between those that occur on the GLYDe Dressing treated side and those that occur on the control side. All available data will be used. No imputation will be performed for missing data for any analysis.
Arm/Group | GLYDe Dressing | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes